CLINICAL TRIAL: NCT05177939
Title: Phase III Study to Evaluate the Efficacy and Safety of NPB-01 in Patients With Autoimmune Encephalitis Refractory to Steroid Pulse Therapy
Brief Title: Phase III Clinical Study of NPB-01 in Patients With Autoimmune Encephalitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPB-01-19/C-01
Record Dates: First submitted 2021-12-03; First posted 2022-01-05 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-01

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Immunoglobulins, Intravenous; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPB-01 (Experimental): Intravenous immunoglobulin
  Interventions: Drug: NPB-01
- NPB-01-ME (Active Comparator): methylprednisolone sodium succinate
  Interventions: Drug: NPB-01-ME

INTERVENTIONS:
Drug: NPB-01 — NPB-01 will be administered for the treatment of autoimmune encephalitis
  Other Names: Intravenous immunoglobulin
  Arms: NPB-01
Drug: NPB-01-ME — NPB-01-ME will be administered for the treatment of autoimmune encephalitis
  Other Names: methylprednisolone sodium succinate
  Arms: NPB-01-ME

SUMMARY:
To compare the efficacy and safety of NPB-01 in patients with autoimmune encephalitis refractory to steroid pulse therapy using steroid pulse therapy as a control.

ELIGIBILITY:
Inclusion Criteria

* < At 1st registration > Patients meeting the possible diagnostic criteria for autoimmune encephalitis
* < At 1st registration > Patients with a CASE score of 5 to 22 during the screening period
* < At 1st registration > Patients with autoimmune encephalitis in progress (active and requiring therapeutic intervention)
* < At 1st registration > IVIG therapy and steroid pulse therapy are considered necessary by the investigator.
* < At 1st registration > Patients aged 15 years or older at the time of informed consent
* < At 2nd registration > Patients who meet any of the following (1) to (6):

  1. Definite diagnostic criteria for autoimmune limbic encephalitis
  2. MRI evidence of demyelination (probable autoimmune encephalitis)
  3. Probabilistic diagnostic criteria for anti-NMDAR encephalitis
  4. Probabilistic diagnostic criteria for Bickerstaff brainstem encephalitis
  5. Probabilistic diagnostic criteria for Hashimoto's encephalopathy
  6. Diagnostic Criteria for Autoimmune Encephalitis with Negative but Probable Autoantibodies
* < At 2nd registration > CASE score of 5 to 22 on Day 8 of the previous treatment period
* < At 2nd registration > Patients who have had an inadequate response to steroid pulse therapy

Exclusion Criteria:

* < At 1st registration > Patients with strongly suspected infectious encephalitis
* < At 1st registration > Patients who received immunoglobulin preparations within 8 weeks prior to informed consent
* < At 1st registration > Patients who received plasma exchange within 4 weeks prior to informed consent
* < At 1st registration > Patients who received immunosuppressants (Rituximab, cyclophosphamide, etc.) within 4 weeks prior to informed consent
* < At 1st registration > Patients who have had tumor resection associated with autoimmune encephalitis within 4 weeks prior to informed consent
* < At 1st registration > Patients with a history of shock or hypersensitivity to the ingredients of NPB-01
* < At 1st registration > Patients with known IgA deficiency
* < At 1st registration > Patients with renal disorder
* < At 1st registration > Patients with a current or previous history of cerebral or cardiovascular disorders (Asymptomatic cerebral infarction and myocardial infarction that occurred more than 5 years ago are not applicable.)
* < At 1st registration > Patients at high risk of thromboembolism
* < At 1st registration > Patients with haemolytic/blood loss anaemia
* < At 1st registration > Immunosuppressed/immunocompromised patients
* < At 1st registration > Patients with decreased cardiac function
* < At 1st registration > Pregnant, expected (desired or planned) pregnant, or breastfeeding patients
* < At 1st registration > Use of prohibited medications or treatment in this study
* < At 1st registration > Patients who received investigational product in this study (re-enrollment prohibited)
* < At 1st registration > Patients who have received treatment with investigational product other than this study within 4 months prior to informed consent
* < At 1st registration > Patients with a history of hypersensitivity to methylprednisolone sodium succinate
* < At 1st registration > Patients who have a tumor associated with autoimmune encephalitis and are considered to require resection during the study period.
* < At 1st registration > Patients receiving intravenous general anesthetics or sedative hypnotics
* < At 1st registration > Patients in coma
* < At 1st registration > Ventilated patients
* < At 1st registration > Patients who cannot undergo protocol-specified tests/assessments
* < At 1st registration > Other patients considered ineligible for the study by the investigator
* < At 2nd registration > Positive herpes simplex virus DNA qualitative test in the screening period.
* < At 2nd registration > Serum creatinine ≥ 2 times the upper limit of normal during the screening period.
* < At 2nd registration > Total protein ≥ 9 g/dL during the screening period.
* < At 2nd registration > Patients with hematocrit ≥ 55% during the screening period
* < At 2nd registration > Patients who meet any of the exclusion criteria at the time of first registration

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders in CASE (Clinical Assessment Scale in Autoimmune Encephalitis) | 4 weeks
  A responder is defined as a patient whose CASE score at Week 4 of the post-treatment follow-up period after treatment with investigational product improved by 40% or more compared to the pre-treatment period.

SECONDARY OUTCOMES:
CASE | 1, 2, 3, 4, 6, 8, 12 weeks
  The change in CASE score at each time point after the start of treatment with investigational product compared with that on Day 8 of the pretreatment period will be compared between the arms. Changes in CASE scores divided into three segments (0 -4: excellent, 5 -9: moderate, 10 -27: poor) will also be compared.
  In addition, the period until CASE score becomes 4 points or less after the start of treatment with investigational product will be checked.
mRS | 1, 2, 3, 4, 6, 8, 12 weeks
  Changes in mRS at each time point after the start of investigational product treatment compared with Day 8 of the pretreatment period will be compared between the arms.
GCS | 1, 2, 3, 4, 6, 8, 12 weeks
  To compare the change in GCS at each time point after the start of investigational product with that on Day 8 of the pretreatment period between the arms.
MMSE-J | 4, 8, 12 weeks
  The change in MMSE-J at each time point after the start of investigational product as compared with Day 8 of the pretreatment period will be compared between the arms.
FAB | 4, 8, 12 weeks
  The change in FAB at each time point after the start of investigational product as compared with Day 8 of the pretreatment period will be compared between the arms.
Disappearance of abnormal EEG findings | 4, 12 weeks
  The proportion of subjects in whom abnormal findings in EEG disappeared at each time point after the start of investigational product as compared with Day 8 of the pretreatment period will be compared between the arms.
Disappearance of abnormal head MRI findings | 4, 12 weeks
  The proportion of subjects in whom abnormal findings in head MRI disappeared at each time point after the start of investigational product as compared with Day 8 of the pretreatment period will be compared between the arms.
Cerebrospinal fluid test | 4, 12 weeks
  The proportion of subjects in whom the cell count returned to within the reference range (≤ 5/μl) and the proportion of subjects in whom the protein count returned to within the reference range (15.0 ~ 45.0 mg/dL) at each time point after the start of investigational product treatment as compared with Day 8 of the pretreatment period will be checked.
Duration of hospitalization | 12 weeks
  Duration of hospitalization after the start of treatment with investigational product to be compared between the arms.
mRS proportion | 1, 2, 3, 4, 6, 8, 12 weeks
  The proportions of subjects with an mRS score of ≤ 2, subjects with an improvement of ≥ 1 point, and subjects with an improvement of ≥ 2 points will also be compared.
  Also, the time to mRS improvement after the start of treatment with investigational product (≤ 2 points, ≥ 1 point improvement, ≥ 2 points improvement) .
GCS proportion | 1, 2, 3, 4, 6, 8, 12 weeks
  Changes in GCS when divided into three segments (15-13: Mild, 12-9: Moderate, 8-3: Severe) will also be compared.
  In addition, the period until the GCS score reaches 13 or higher after the start of treatment with investigational product will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Mamoru Ota, Study Chair — Nihon Pharmaceutical Co., Ltd
Locations (1):
- Trial site 1, Ube, Yamaguchi, Japan